CLINICAL TRIAL: NCT05480644
Title: Circulating Biomarkers Repository in Adults Diagnosed With Primary and Metastatic Brain Tumors
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110602
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor, Primary; Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma for circulating tumor DNA analysis Whole blood for peripheral blood mononuclear cell and circulating immune cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this protocol is to create a repository of blood samples from patients diagnosed with primary and metastatic brain tumors who are being seen in the Department of Radiation Oncology at Duke Cancer Center.

DETAILED DESCRIPTION:
Repository blood samples will be used to study the association of circulating biomarkers with radiation therapy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of primary or metastatic brain tumor (histology or imaging as appropriate)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary or metastatic brain tumors and treated in the Department of Radiation Oncology at Duke
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Number of circulating immune cells in peripheral blood | 6 weeks post radiation therapy
  reported as mean +/- standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Vaios, MD MBA, Principal Investigator — Duke University Health System (DUHS)
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No